CLINICAL TRIAL: NCT01698528
Title: Evaluation of a Prototype Diabetes Management System Applied to Insulin Initiation and Titration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Massachusetts Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHS 2012-18
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Results first posted 2017-09-14 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-09

CONDITIONS: Type II Diabetes
Keywords: Diabetes; diabetes technologies; telemedicine
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): The experimental arm will be provided with a tablet computer with a newly designed software to help manage his or her diabetes care. This arm will communicate with his or her provider through the tablet computer to initiate and titrate basal insulin dose based on the 303 protocol. The individuals in this arm will also track their glucose values and medication adherence using the tablet computer by documenting when medication was taken or insulin was injected.
  Interventions: Device: Tablet Computer
- Control Group (No Intervention): The individuals in the control group will receive usual care from the study Clinic as they always have. These individuals will be tracking their diabetes in the same way they have been by communicating with their health care provider and his or her office via fax/phone/e-mail. These individuals will not be provided with a tablet computer.

INTERVENTIONS:
Device: Tablet Computer
  Other Names: Toshiba tablet computer
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to determine if using a diabetes management technology system, including a tablet computer, to track diabetes care and communicate with a clinician coach (a doctor or nurse from the Joslin Clinic) makes starting and adjusting insulin easier and safer for people with type 2 diabetes. Hypothesis: The use of a diabetes management technology system with a clinician coach helps more individuals starting basal insulin achieve better glycemic control with less hypoglycemia compared with standard clinical practice at Joslin Diabetes Center.

ELIGIBILITY:
Inclusion:

* 18 years or older
* Has type 2 diabetes, starting on basal insulin therapy
* Hemoglobin A1c between 9-14%
* Has Wi-Fi internet connection at home
* Is willing to monitor blood glucose at least once per day
* Is willing to inject and self-titrate insulin dose
* Able to read and communicate in English proficiently

Exclusion:

* Has severe visual impairment impacting visual acuity
* Has severe hearing impairment impacting communication
* Has Type 1 diabetes
* Pregnant or lactating women
* Alcohol dependency
* Require multiple daily insulin injections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Hsu, M.D., Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: The experimental arm will be provided with a tablet computer with a newly designed software to help manage his or her diabetes care. This arm will communicate with his or her provider through the tablet computer to initiate and titrate basal insulin dose based on the 303 protocol. The individuals in this arm will also track their glucose values and medication adherence using the tablet computer by documenting when medication was taken or insulin was injected.
  Tablet Computer
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 20 | 20
Completed | 19 | 16
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (16.04) | 53.3 (1.88) | 53.52 (13.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 13 | 13 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Control as Determined by the Change in Absolute HbA1c Level
Description: The primary outcome of interest is absolute decrease in A1c by end of 3 months.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Percent A1C
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
Percent A1C | -3.16 (1.54) | -2.00 (2.03)

2. Secondary Outcome: Number of Participants Reaching Target of HbA1c ≤ 7%
Description: Secondary outcomes will include % of participants reaching glycemic target of A1c≤7.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
Participants | 8 | 5

3. Secondary Outcome: Change in Average Participation Satisfaction
Description: The volunteer's satisfaction with their diabetes care will be measured at the beginning and at the end of the study. Diabetes Treatment Satisfaction Questionnaire (DTSQ) was used for assessing the satisfactory level. DTSQ consisted of 8 questions, each question with a score scale of 0-6 (very dissatisfied to very satisfied), leading to a final score range of 0-48, with higher scores indicating greater satisfaction. The change in the DTSQ comparing before (time 0) and end of the study (t=3months) was measured. The average change in the intervention group and control group were listed in the outcome measure data table.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
Scores on a scale | 10.1 (11.68) | 2.05 (6.45)

4. Secondary Outcome: Number of Participants With Hypoglycemia
Description: Number of participants had hypoglycemia during the trial period
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
Participants | 3 | 1

5. Secondary Outcome: Time Health Care Providers and Subjects Spend on Managing the Insulin Titration
Description: time health care providers and subjects spend on managing the insulin titration through appointment, phone call, emails, faxes
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
min | 108 (41) | 80 (51)

ADVERSE EVENTS:
Arm/Group | Intervention Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes